CLINICAL TRIAL: NCT06928077
Title: Inspiration From Eye-tracking Data: Investigating the Impact of Combining Specific Environmental Features and Power Mobility Training on Functional Skills and Caregiver-child Interaction in Toddlers With Motor Delays
Brief Title: Inspiration From Eye-tracking Data: Investigating the Impact of Combining Specific Environmental Features and Power Mobility Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiang-Han Huang, Associate Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 113WFD2610113
Record Dates: First submitted 2025-03-29; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Young Children With Motor Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ROC-Stand training with specific environmental features (ROC-Stand(SE)) (Active Comparator): Each session will last for 2 hours, occurring twice a week over a 12-week intervention period, and will be based on ecological and dynamic systems theories.Weekly, the research team will assist participants in wearing a lightweight HMET to record the first 10 minutes of both the driving and natural play sessions during each 2-hour training session. This will result in a total dataset of 20 minutes per session. Each training session structure includes a 70-minute driving session and a 40-to-50-minute natural play session, with an optional 10-minute break, as needed, in line with ROC-related studies. These discussions and coaching methods will also be informed by clinical observations of the participant's performance in prior sessions.
  Interventions: Behavioral: ROC-Stand training with specific environmental features
- ROC-Stand training without specific environmental features (ROC-Stand(NSE)) (Active Comparator): The same therapist responsible for the ROC-Stand(NSE) group will oversee the program. This group's training frequency will match that of the ROC-Stand(SE) group, adhering to training principles similar to those employed in previous ROC training studies in various environments. Furthermore, during each training session, participants will wear the HMET for 20 minutes, capturing the initial 10 minutes of both the driving and natural play segments.
  Interventions: Behavioral: ROC-Stand training without specific environmental features
- Conventional therapy (Control) (Active Comparator): The frequency and duration of these sessions are identical to those in the ROC training groups, with objectives tailored to enhance specific motor or psychosocial skills relevant to each participant's current developmental stage. They will also wear the HMET for the first 20 minutes of one training session each week, enabling the collection of similar data to that gathered from the ROC training groups.
  Interventions: Behavioral: Conventional therapy

INTERVENTIONS:
Behavioral: ROC-Stand training with specific environmental features — A licensed, independent therapist along with caregivers will conduct the training program in a public space at the university. The initial phase of the training will concentrate on developing the participants' understanding of cause-and-effect in relation to the control system and the movement of the car, focusing on specific public spaces such as hallways, convenience stores, gardens, and museums. Following this, the therapist will collaborate with caregivers to direct the participants' gaze towards specific physical structures and objects. Furthermore, the therapist will guide and coach caregivers on how to lead the participants in engaging with these environmental features through various exploratory actions, as supported by previous evidence. These actions include touching, hitting, squeezing, pointing, holding objects with one or two hands, object touching own body, fingering, banging, manipulating, and transferring objects.
  Arms: ROC-Stand training with specific environmental features (ROC-Stand(SE))
Behavioral: ROC-Stand training without specific environmental features — The initial phase of training will also focus on teaching participants about cause-and-effect as it pertains to the control system and movement of the car. This phase will include goal-oriented driving activities, such as traveling 200 meters to reach a preferred toy or to interact with someone, and engaging in games like hide-and-seek in various public spaces including hallways, convenience stores, gardens, and museums. The training, without a specific emphasis on environmental features, will highlight the use of upper limbs in functional tasks during driving sessions, and incorporate a range of motor skills to enhance mobility and socialization during natural play sessions. The details of the program will also be established through collaborative discussions between the family and the treating therapist. These discussions will take into account clinical observations of the participant's performance in previous sessions.
  Arms: ROC-Stand training without specific environmental features (ROC-Stand(NSE))
Behavioral: Conventional therapy — The overarching goal of this training is to support developmental progress and improve mobility, socialization, and upper limb functionality in everyday tasks. Participants in this group will have the opportunity to walk in the same public space used by the ROC training groups, allowing interaction with both the therapist and caregivers based on their individual motor capabilities.
  Arms: Conventional therapy (Control)

SUMMARY:
This study has three main objectives. First, the investigators want to see how using a lightweight head-mounted eye tracker (HMET) can help to understand looking behavior, visual focus, and social interaction in toddlers with motor delays during ROC-Stand training. The investigators will compare the effects of training with specific environmental features to training without these features and to conventional therapy. Second, the investigators will evaluate outcomes related to body function, daily activities, and participation, along with family perceptions and involvement, using the ICF framework. Third, the investigators will explore how temperament, motivation, looking behavior, and caregiver-child interactions relate to each other in these toddlers across different training programs.

Based on previous research, the investigators plan to recruit 30 toddlers with motor delays and randomly assign them to one of three groups: ROC-Stand with specific environmental features (ROC-Stand(SE)), ROC-Stand without these features (ROC-Stand(NSE)), and conventional therapy (Control), with 10 toddlers in each group. Each toddler will receive a total of 48 hours of training over 24 weeks, with two 120-minute sessions per week-12 weeks of intervention followed by a 12-week follow-up. The participants will also continue their regular therapy during the study. The HMET will record visual and manual behaviors for 20 minutes each week, and standardized assessments of body function, mobility, psychosocial function, family perception, and participation will be done before the intervention, after the intervention, and at the end of the follow-up.

The findings from this study will help identify key environmental factors for early power mobility training and provide families and therapists with a clear, structured approach to using these techniques.

DETAILED DESCRIPTION:
Environmental and task modifications are widely used in pediatric rehabilitation to help shape children's actions. However, therapists often adjust these factors by trial and error. A better understanding of how to optimize the "fit" between a child and their surroundings could lead to a more systematic approach, making it easier for children to develop new actions. Head-mounted eye trackers (HMETs) are wearable devices that record eye movements in real-world settings. By combining ROC (ride-on car) training with HMET technology, the investigators can track the visual and touch-based information that young children gather as they use power mobility devices (PMDs). This new approach helps to see how toddlers interact with their environment, deepening our understanding of their development.

This research project focuses on three key aims: 1) Evaluating the effects of ROC-Stand training programs, both with and without specific environmental features, on the looking behaviors and social interactions of toddlers with motor delays, compared to a control group receiving conventional therapy; 2) Determining the effectiveness of these programs in achieving various outcomes as categorized by the International Classification of Disability, Functioning, and Health (ICF) framework for toddlers with motor delays; and 3) Investigating how these training programs affect the relationship among children's temperament, mastery motivation, looking behaviors, and caregiver-child interactions in toddlers with motor delays.

Study design: The investigators will use a randomized, pretest-posttest control group design with three groups. The study will involve a three group comparison: two ROC training programs, differentiated by the inclusion (ROC-Stand(SE)) or exclusion (ROC-Stand(NSE)), of specific environmental features, and a control group receiving conventional therapy. All groups will have an identical training schedule: 2-hour sessions, conducted twice a week for a 12-week period. The duration of the study for each participant is set at 6 months, which includes a 3-month intervention period followed by a 3- month follow-up phase. Participants will continue their regular therapy sessions throughout the study.

Participants: The study will include 30 toddlers, aged between 12 to 36 months, who have motor delays. These participants will be randomly assigned into three groups, each consisting of 10 toddlers: the ROC-Stand(SE) group, the ROC-Stand(NSE) group, or the Control group. The sample size for our study on early powered mobility training is determined based on an effect size (f) of 0.3, as observed in a previous ROC-Stand RCT that assessed social function in PEDI-C. This calculation takes into account a statistical power of 0.8, a two-sided type I error rate of 0.05, an anticipated dropout rate between 20 to 25%, and recruitment conditions from prior studies.

Recruitment: Participants will be recruited through self-referrals, healthcare practitioners, and hospitals in Taoyuan or New Taipei where toddlers receive outpatient rehabilitation. Flyers will be distributed in clinical settings, and interested parents will be contacted to explain the study details. Informed consent will be obtained before enrollment.

Procedure: Before the intervention, toy cars will be modified for safety-seats will be adjusted and the acceleration system changed to a switch. Toddlers in the ROC training groups will receive these custom-made, standing-style cars. Pre-intervention assessments will be conducted by an independent occupational therapist who is unaware of the study's goals and group assignments. These assessments, carried out in a testing room at Chang Gung University, will occur at three time points: before training (T1), three months into training (T2), and three months after training ends (T3). The assessments will take place in a testing room at Chang Gung University, occurring at three different times: before training (T1), three months after the start of the training (T2), and three months following the end of the training (T3). All participants will begin their respective training programs at the university. During the intervention, each toddler will wear a lightweight HMET for 20 minutes once a week to record eye gaze, manual actions, and social interactions. An activity log will document the training conditions and capture caregivers' weekly feedback. In the follow-up phase, participants will not receive any training from our research team. Instead, they will continue with their regular therapy at their clinics. We will gather information about this regular therapy, including its type, frequency, and dosage, at three time points: T1, T2, and T3. All eye-tracking data will be analyzed by two independent coders, who are undergraduate students. Before they begin their analysis, the principal investigator (PI) will instruct them on coding procedures. To ensure reliability, Cohen's kappa coefficient will be calculated between the two raters before formal coding.

Intervention (training phase): One licensed occupational therapist who is responsible for providing the training programs, will collaborate with caregivers to set goals and track progress using goal attainment scaling (GAS) at T1, T2, and T3 for all three groups. These goals will pertain to aspects of mobility and psychosocial functions. The ROC-related training programs will involve one therapist working closely with the caregivers, employing coaching techniques from the FCS model. Furthermore, the programs incorporate a standing posture and are context-focused. The conventional therapy program, on the other hand, is a child-centered, therapist-directed approach. Participants will be allowed necessary breaks during training sessions based on their endurance. In addition, all participants in the three groups will wear a lightweight HMET (weighing 46 g) from Positive Science, LLC to record their looking, fixation, and interactive behaviors during one session per week of the intervention. All participants will continue their regular therapy (e.g., physical, occupational, speech therapy) throughout the 6-month study.

Follow-up: During this period, a follow-up phase will take place after the completion of the training programs mentioned above. In this phase, participants will not receive any additional training programs from the study but will continue with their regular therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 1 to 3 years
2. having motor delays that either prevent independent walking or require the use of assistive technology for walking, defined as more than 1.5 standard deviations(SD) below the mean, as evaluated by the Chinese Child Development Inventory via a physician
3. able to stand independently for at least two seconds or can tolerate standing with support for up to 10 minutes
4. capable of reaching for objects with either one or both hands
5. with a height ranging from 69 to 103 cm and a weight between 7 to 18 kg
6. having parents who can provide consent for their child's participation in the training programs

Exclusion Criteria:

1. children with severe sensory impairments, such as blindness or deafness
2. children whose height falls outside the range of 69 to 103 cm and weight outside the range of 7 to 18 kg
3. parents or caregivers who are unable to commit the time required for the training phase
4. children who exhibit severe emotional reactions that could potentially lead to harm

Ages: 10 Months to 40 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Looking Behaviors, Visual Fixation, and Social Interactions Assessed Using the Positive Science Head-Mounted Eye Tracker (HMET) | Once per week during the intervention phase, for a 20-minute session (weekly for 12 weeks)
  Participants' visual behaviors and social interactions will be assessed weekly during the training phase using the Positive Science Head-Mounted Eye Tracker (HMET). This objective eye-tracking system includes a 46 g lightweight headgear, a cap, wireless transmitter, and battery pack (total weight 271 g). An infrared eye camera tracks the participant's right eye movements, and a forward-facing scene camera captures the environment with a 90° field of view.
  Live Capture software (Positive Science) records synchronized eye and scene videos at 30 Hz. Eye-tracking calibration is conducted using Yarbus software (Positive Science), which generates gaze point visualizations with a 4° radius marker on each video frame. A trained therapist monitors recordings in real time.
  Each participant will be recorded for 20 minutes per week during the training period. Videos will be coded offline using a protocol adapted from established infant research. Coded behaviors include looking at faces, bodies,

SECONDARY OUTCOMES:
The Bayley Scales of Infant and Toddler Development-Third Edition (Bayley-III) | The test will be administered on three occasions: before and after the 3-month intervention (T1 & T2) and the end of the 3-month follow up phase (T3).
  An internationally recognized set of developmental tests with high reliability and validity applied to examine participants' developmental abilities. The Bayley has subsets of tests for motor, cognitive, and language development for children aged from 1 month to 42 months. It is a standardized assessment that can classify children's severity level of motor delays into four levels based on their motor composite scores, classified as severe (scores <55), moderate (55-69), mild (70-84), and no (>85) motor delays.
Toddler Temperament Scale (TTS) | The test will be administered on three occasions: before and after the 3-month intervention (T1 & T2) and the end of the 3-month follow up phase (T3).
  A standardized tool designed to assess temperamental characteristics in children aged 1 to 3 years. Caregivers are given statements describing specific behaviors and are asked to rate the frequency of these behaviors in their child using a 6-point scale. The scoring of the results is structured such that higher scores correspond to a more challenging temperament.
Peabody Developmental Motor Scales - Third edition (PDMS-3) | The test will be administered on three occasions: before and after the 3-month intervention (T1 & T2) and the end of the 3-month follow up phase (T3).
  A norm-referenced, standardized tool for assessing gross and fine motor skills in children from birth up to 5 years and 11 months.This assessment comprises five core subtests and one supplemental subtest, which evaluate body control, body transport, object control, hand manipulation, eye-hand coordination, and physical fitness.
The Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version | The test will be administered on three occasions: before and after the 3-month intervention (T1 & T2) and the end of the 3-month follow up phase (T3).
  A caregiverreported tool using a five-point scale to measure both instrumental and expressive aspects of mastery motivation. Comprising seven subscales, the DMQ evaluates cognitive/object persistence, gross motor persistence, social mastery motivation with adults, social mastery motivation with children/peers, mastery pleasure, reactions to challenge in mastery situations, and general competence. A higher DMQ score is indicative of greater motivation. For children aged 6 months to 19 years, the DMQ 18 previously showed good validity and reliability. Considering the age of participants, this study used two versions of the DMQ 18: infant's version (6-18 months) and preschooler's version (1.5-5 years).
The Chinese version of Pediatric Evaluation of Disability Inventory (PEDI-C) | The test will be administered on three occasions: before and after the 3-month intervention (T1 & T2) and the end of the 3-month follow up phase (T3).
  A comprehensive set of assessments designed for children aged 8 months to 6 years. It effectively quantifies self-care, mobility, and social function, making it particularly valuable for monitoring changes in functional skills. Each domain within the PEDI-C can be analyzed independently. The study has demonstrated excellent inter-rater and intra-rater reliabilities, showing high consistency in observations (ranging from 0.95 to 0.99), and good concurrent validity when compared with the Functional Independence Measure for Children, as indicated by Spearman correlation coefficients ranging from 0.92 to 0.99.
Goal Attainment Scale (GAS) | The test will be administered on three occasions: before and after the 3-month intervention (T1 & T2) and the end of the 3-month follow up phase (T3).
  A family-centered, criteria-referenced, responsive tool that includes five possible outcomes. A score of 0 signifies that the child has achieved the specified goal. Scores of -2 and -1 indicate performance levels below expectations, while +1 and +2 reflect performance that exceeds expectations. This tool has demonstrated good validity and excellent inter-rater agreement, with Intraclass Correlation Coefficients (ICCs) of 0.90 or higher. The individual goals are incorporated into a single GAS composite score, which is then converted into a T-score. A mean Tscore of 50 suggests that participants have exceeded the anticipated level of goal achievement.
The Chinese version of the Affordance in the Home Environment for Motor Development - Toddler version (AHEMD-Toddler-C) | The test will be administered on three occasions: before and after the 3-month intervention (T1 & T2) and the end of the 3-month follow up phase (T3).
  A reliable and valid tool for evaluating the quality and quantity of motor development opportunities available in the home environment during early childhood. 72 Age-specific AHEMD questionnaires have been developed for different age ranges: 3-to-18 months and 18-to-42 months. These questionnaires have been translated into Chinese. The test-retest reliabilities for the AHEMD-Toddler-C are adequate, ranging from 0.46 to 0.93. Regarding convergent validity, the correlation coefficients between the AHEMD and the Home Observation for Measurement of the Environment (HOME) inventory stand at 0.44.
The Parenting Stress Index Short Form (PSI/SF) | The test will be administered on three occasions: before and after the 3-month intervention (T1 & T2) and the end of the 3-month follow up phase (T3).
  A tool to assess the overall level of parenting stress experienced by parents or caregivers of children aged between one month and 12 years. It comprises three subscales: parental distress, parent-child dysfunctional interaction, and difficult child, which collectively contribute to a total stress score. A higher score on this scale signifies increased stress levels. Known as the PSI/SF, this tool is recognized for its excellent validity and reliability.
Activity Log | The test will be administered on three occasions: before and after the 3-month intervention (T1 & T2) and the end of the 3-month follow up phase (T3).
  To document the training duration, locations, activities, and the caregiver's feedback on the training program weekly during the intervention phase. This log will primarily consist of qualitative data, including detailed descriptions provided by parents.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Han Huang, ScD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan, Taoyuan County, Taiwan